CLINICAL TRIAL: NCT04081142
Title: Application of Indicator Based-EIT Method Assess Lung Regional Perfusion for Critically Ill Patients in ICU
Brief Title: Application of Indicator Based-electrical Impedance Tomography Method Assess Lung Regional Perfusion in ICU Patients
Status: Completed | Type: Observational
Sponsor: Yun Long (Other)
Responsible Party: Sponsor-Investigator, Yun Long, the director of the intensive care medicine, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: EIT-lung Perfusion in ICU
Record Dates: First submitted 2019-09-03; First posted 2019-09-09 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Respiratory Failure; Hypoxemia; ARDS, Human
Keywords: EIT, pulmonary perfusion
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- acute respiratory failure group: acute respiratory failure (ARF) group: arterial oxygen partial pressure to fractional inspired oxygen ratio, PaO2/FiO2<300 mmHg and/or peripheral oxygen saturation SaO2<94% under air condition and/or severe dyspnea with respiratory rate >30bpm.
- control group: postoperative ICU patients without ARF were included

SUMMARY:
This study is an observational study. Investigate the relationship of oxgenation and lung regional ventilation and perfusion assessed by the indicator based-EIT method in the critically ill patients in ICU

DETAILED DESCRIPTION:
1. Written informed consent was obtained from all patients or next of kin before data were included in the study.
2. When the research team was available, adult patients within 1w, who were sequentially admitted to the Department of Critical Care Medicine and required central venous catheters for resuscitation were eligible for the study.
3. Information collected at enrollment included demographic characteristics such as age, sex, Acute Physiology and Chronic Health Evaluation II score (APCHEII); . The global hemodynamic, respiration condition and PaO2 were measured. At the same time, the lung regional ventilation and perfusion assessed by the indicator based-EIT method(injection 10%NaCL).
4. The 10%NaCL was injected by the central venous catheter.

ELIGIBILITY:
Inclusion Criteria:

* Time of admission ICU < 7days
* Age (> 18 years old)
* Have been placed central venous catheter based on clinical requirement

Exclusion Criteria:

.Chest skin injured and cannot be monitored by EIT.

* Severe Hypernatremia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients within 7days, who were sequentially admitted to the Department of Critical Care Medicine and required central venous catheters for clinical requirment were eligible for the study.
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Lung regional perfusion | Hour 1
  Lung regional perfusion monitored by EIT with saline
oxygenation | Hour 1
  oxygenation(SpO2) measured by bedside monitor

CONTACTS AND LOCATIONS:
Overall Officials: Yun Long, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang Q, Su L, Jiang J, Wang N, He H, Long Y. Incorporating electrical impedance tomography to transpulmonary pressure-guided PEEP in severe ARDS with pneumothorax and multiple cavitations: a case report. Front Med (Lausanne). 2023 Aug 28;10:1240321. doi: 10.3389/fmed.2023.1240321. eCollection 2023. PMID 37700773
- [Derived] He H, Chi Y, Long Y, Yuan S, Zhang R, Yang Y, Frerichs I, Moller K, Fu F, Zhao Z. Three broad classifications of acute respiratory failure etiologies based on regional ventilation and perfusion by electrical impedance tomography: a hypothesis-generating study. Ann Intensive Care. 2021 Aug 28;11(1):134. doi: 10.1186/s13613-021-00921-6. PMID 34453622